CLINICAL TRIAL: NCT01132261
Title: A Randonized Control Trial of a Brain Preservation Diet in Preventing Congnitive Decline in Odl Age Hostel Residents
Brief Title: Trial of a Brain Preservation Diet in Preventing Cognitive Decline in Old Age Hostel Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Professsor, Thhe Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCT-dietetic intake; CRE-2005.473
Record Dates: First submitted 2010-05-25; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-01

CONDITIONS: Cognitive Decline; Dietetic Intake
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): brain preservation diet
  Interventions: Other: "brain preservation' diet
- 2 (No Intervention)

INTERVENTIONS:
Other: "brain preservation' diet — dietetic evaluation and advice in small group for health diet
  Arms: 1

SUMMARY:
Dementia is a major cause of disabilities in older people. If the onset of dementia can be delayed by preventive measures, the burden of the disease to the society can be greatly reduced. It is now recognised that dietary factors are related to the incidence of dementia. High intake of vegetables, fruit and fish are protective while high intake of saturated fat and salt (via its effect on blood pressure) are detrimental to risk of dementia.

The investigators therefore propose to perform a randomized controlled trial of dietetic interventions in old age hostels in Hong Kong. Twelve old age hostels under the Tung Wah Group will be randomly assigned to intervention or control groups. The intervention group will receive dietetic interventions by 2 weekly small group discussion with the residents, modification of menu and publicity. The daily diet to be implemented consists of the following principles: 1. fresh fruit 2 portions, 2. vegetables 4 portions, 3. fish, 4. white meat, 5. sodium intake < 100 mmol/L, 6. six glasses of water. In the control group. The dietician will give two health talks and advice on menu only.

The primary outcome is the incidence of questionable dementia in those who are normal at baseline and the incidence of dementia in those who have questionable dementia at baseline. The categorisation will be performed by trained research assistant after administering a structured questionnaire. Change in mini-mental examination score and SF36 quality of life scores are secondary outcomes. Food records over three days for each subject are recorded every three months, to ensure that the brain preservation diet has been adhered to. Half of the subjects will be randomly assigned to have blood and urine tests at baseline and at one year, in order to examine the health effects of dieting.

ELIGIBILITY:
Inclusion Criteria:

* old age home residents age 75 years or above, CDR<1

Exclusion Criteria:

* tube fed residents

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
cognitive decline | 33 months

SECONDARY OUTCOMES:
Change in MMSE test | 33 months
% subjects meeting targets of brain preservation diet | 33 months
  brain preservation diet includes 3 portion of vergetables per day, 2 portion of fruit per day, 5 meal of fish per week, 6 glasses of water per day.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Kwok TC, Lam LC, Sea MM, Goggins W, Woo J. A randomized controlled trial of dietetic interventions to prevent cognitive decline in old age hostel residents. Eur J Clin Nutr. 2012 Oct;66(10):1135-40. doi: 10.1038/ejcn.2012.117. Epub 2012 Sep 5. PMID 22948946